CLINICAL TRIAL: NCT01386827
Title: Ability of the New Vero-cell-derived Inactivated Japanese Encephalitis Vaccine (IXIARO) to Elicit a Booster Response in Travellers Previously Vaccinated With Traditional Mouse-brain Derived Vaccine (JE-MB)
Brief Title: Ixiaro as Booster After Mouse-brain Derived Vaccines for Japanese Encephalitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anu Kantele, Associate professor, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 382/E7/07
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Japanese Encephalitis
Keywords: Ixiaro; japanese encephalitis vaccine; booster
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Immunization, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A) primary immunization with MB-JEV (Active Comparator): Volunteers immunized with MB-JEV
  Interventions: Biological: Mouse brain derived japanese encephalitis vaccine (MB-JEV)
- Primary and booster MBJEV vaccinations (Active Comparator): Booster immunization with MB-JEV of vaccinees primed with MB-JEV
  Interventions: Biological: Primary and booster immunizations with MB-JEV
- C) primary immunizations with Ixiaro (Active Comparator): Primary immunization with Ixiaro 2 dose
  Interventions: Biological: C) primary immunizations with Ixiaro
- S) Ixiaro booster to MBJEV primed (Active Comparator): Actual study group:Booster immunization with Ixiaro to those primed previously with MB-JEV
  Interventions: Biological: S) Ixiaro booster to MBJEV primed

INTERVENTIONS:
Biological: Mouse brain derived japanese encephalitis vaccine (MB-JEV) — a) 2-3 doses of MB-JEV vaccine 0.5ml given on day 0, 7, 30 immunization and one booster dose of Ixiaro 0.5 ml > 2 years later
  Other Names: Korean Green Cross
  Arms: A) primary immunization with MB-JEV
Biological: Primary and booster immunizations with MB-JEV — 2-3 doses of MB-JEV vaccine 0.5ml given on day 0, 7, 30 as primary immunization and one booster dose of 0.5 ml > 2 years later
  Other Names: Korean Green Cross
  Arms: Primary and booster MBJEV vaccinations
Biological: C) primary immunizations with Ixiaro — 2 0.5 ml doses of Ixiaro 28 days apart
  Other Names: Ixiaro
  Arms: C) primary immunizations with Ixiaro
Biological: S) Ixiaro booster to MBJEV primed — 0.5ml Ixiaro to volunteers previously primed with 2-3 doses of MB-JEV
  Other Names: Ixiaro
  Arms: S) Ixiaro booster to MBJEV primed

SUMMARY:
The old mouse brain derived Japanese encephalitis vaccines (MBJEV) have been reported to cause serious adverse effects and are therefore replaced with the novel Ixiaro vaccine. The present study investigates whether vaccinees primed with MBJEV can be boosted with Ixiaro.

Travellers receiving Japanese encephalitis vaccines are enrolled for a follow-up of immune responses in four groups: A) primary immunization with BMJEV, B) primary and secondary immunizations with MBJEV, C) primary immunizations with Ixiaro and S) Primary immunization with MBJEV and secondary immunization with Ixiaro. Immune responses are followed with help of serum samples collected before and after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Male and female travellers ≥ 18 years of age.

  * General good health.
  * Written informed consent.
  * Ability to attend all visits scheduled in this study.
  * Travellers who have previously got a primary vaccination series of 2 or 3 doses of JE-MB and now receive a booster vaccination , either MB-JEV or IXIARO, at the travel clinic for their journey to Asia, OR
  * Travellers with no previous vaccination against JE who are given the primary vaccination series with IXIARO at a travel clinic prior to their journey to Asia.

Exclusion Criteria:

* - < 18 years of age.
* Acute disease at the time of enrollment.
* Pregnancy or lactation.
* Known immunodeficiency or immune suppressive treatment.
* Any chronic illness that might interfere with the immune response; history of JE.
* Alcohol or drug abuse.
* Any clinically significant history of known or suspected anaphylaxis or hypersensitivity (based on the investigator's judgement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Antibody titers 1 month after last vaccine dose | 1 month
  Determination of antibody titers 1 month after last vaccine dose

SECONDARY OUTCOMES:
Antibody titers two years after vaccination | 2 years
  Measurement of antibody titers two years after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Elina Erra, MD, Principal Investigator — Haartman Institute, University of Helsinki; Lars Lindqvist, MD PhD, Principal Investigator — Department of infectious diseases Stockholm, Sweden; Eili Huhtamo, PhD, Principal Investigator — Haartman Institute, University of Helsinki; Olli Vapalahti, MD PhD, Principal Investigator — Haartman Institute, University of Helsinki; Sari Pakkanen, MSc, Principal Investigator — Haartman Institute, University of Helsinki; Sirkka Vene, BMA, Principal Investigator — Swedish Institute of Infectious Disease Control; Jukka Riutta, MD, Principal Investigator — Travel clinic, Postitalo, Lääkärikeskus; Anu Kantele, MD PhD, Study Director — Helsinki University Central Hospital; Lars Rombo, MD PhD, Study Director — Karolinska Institutet

REFERENCES:
- [Derived] Erra EO, Askling HH, Rombo L, Riutta J, Vene S, Yoksan S, Lindquist L, Pakkanen SH, Huhtamo E, Vapalahti O, Kantele A. A single dose of vero cell-derived Japanese encephalitis (JE) vaccine (Ixiaro) effectively boosts immunity in travelers primed with mouse brain-derived JE vaccines. Clin Infect Dis. 2012 Sep;55(6):825-34. doi: 10.1093/cid/cis542. Epub 2012 Jun 13. PMID 22696017